CLINICAL TRIAL: NCT04285242
Title: Metabolic and Immunological Phenotyping in Patients With Cancer
Acronym: MIPPaC
Status: Recruiting | Type: Observational
Sponsor: CCTU- Cancer Theme (Other)
Responsible Party: Sponsor-Investigator, CCTU- Cancer Theme, Cambridge Clinical Trials Unit - Cancer Theme, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Other Study IDs: MIPPaC
Record Dates: First submitted 2020-02-19; First posted 2020-02-26 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Cancer; Non-Hematologic Malignancy
Keywords: Cancer; Non-haematological
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Participants with Cancer - Group A: Assessments and observations for up to 40 days with one overnight hospital stay.
  Interventions: Other: Observational assessments
- Healthy Volunteers - Group A: Assessments and observations for up to 2 days with one overnight hospital stay.
  Interventions: Other: Observational assessments
- Healthy Volunteers - Group B: Assessments and observations for up to 2 days.
  Interventions: Other: Observational assessments
- Participants with Cancer - Group B: Assessments and observations for up to 40 days, with most assessments and observations being optional and no overnight hospital stay.
  Interventions: Other: Observational assessments

INTERVENTIONS:
Other: Observational assessments — Clinical assessments

SUMMARY:
An observational study to investigate cachexia in participants with non-haematological cancer.

DETAILED DESCRIPTION:
A single-centre, non-randomised, observational study. This study will investigate the systemic metabolic and immunological changes that occur in cachexia. The aim is to better understand the mechanism(s) underlying weight loss in people with non-haematological cancer. This will help to facilitate future research to generate treatments to reverse weight loss and improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent to participate
* Be aged 18 years or over at the time of signing the informed consent form
* Have a histological or cytological diagnosis of a non-haematological cancer
* Are willing and able to comply with study procedures and visits

Exclusion Criteria:

* Active infection, as determined by the investigator based on clinical symptoms and / or fever and / or requirement for antibiotics
* Current treatment with chemotherapy, oral steroids or other immunosuppressive drugs (within 7 days of baseline investigations or during the study phase)
* Significant acute, chronic or psychiatric condition or laboratory abnormality which in the judgment of the investigator would place the patient at undue risk or interfere with the study.
* Intolerance to dairy products
* Women, who are pregnant, plan to become pregnant or are lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and Female participants who have cancer or are healthy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Serum cortisol level | Change from baseline serum cortisol level at Day 2
  Blood serum cortisol levels in weight losing and weight stable patients at baseline and Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Claire Connell, Principal Investigator — University of Cambridge
Locations (2):
- United Kingdom (2):
  - Addenbrooke's Hospital, Cambridge University Hospitals Foundation Trust,, Cambridge, Cambridgeshire
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge, England

IPD SHARING:
Plan to Share IPD: No